CLINICAL TRIAL: NCT05761535
Title: Big Data and Genomic Imaging for the Development of Biomarkers and Nanovector Drugs Innovative for Diagnosis and Therapy of Inflammatory Processes in Dementia
Acronym: BigImAGING
Status: Completed | Type: Observational
Sponsor: IRCCS SYNLAB SDN (Other)
Responsible Party: Sponsor
Other Study IDs: 6/20
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-02

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neurological disease patients: 150 patients with Alzheimer's disease (AD) and Parkinson's disease (PD) for MRI and PET examinations and laboratory medicine
  Interventions: Radiation: Magnetic Resonance (MR) and positron emission tomograph (PET) imaging analyses
- healthy subjects: Healthy subjects
  Interventions: Radiation: Magnetic Resonance (MR) and positron emission tomograph (PET) imaging analyses

INTERVENTIONS:
Radiation: Magnetic Resonance (MR) and positron emission tomograph (PET) imaging analyses — Regarding the neurological MR protocol, the following may be acquired:
  * 3D T1 and T2 high-resolution sequences, acquired in a specific plane and Multiplanar reformation (MPR) reconstructed in the remaining orthogonal planes, for morphological assessment of the different structures under examination;
  * diffusion sequences for the evaluation of the connection between different areas within a specific organ;
  * perfusion sequences (ASL, arterial spin labeling) for the evaluation of perfusion without ev mdc administration;
  * susceptibility sequences for noninvasive assessment of vasculature and deposits of iron.

SUMMARY:
The correlation between data obtained by "imaging" in patients with neurodegenerative diseases characterized by inflammation and the presence in the peripheral blood of the same patients "biopsies liquid biopsies" of specific circulating nucleic acids, could enable the development of methods and algorithms capable of identifying novel biomarkers that serve as targets for the development of probes diagnostics and therapeutics. This is the context for the project idea, which is aimed at developing development of a performant multi parameter system capable of identifying novel biomarkers of microglial polarization that can be used for diagnostic and prognostic purposes in determining the staging/progression of neurodegenerative disease

ELIGIBILITY:
Inclusion Criteria:

All subjects of either sex aged 18 to 85 years who are able to provide voluntary consent, suffering from neurodegenerative diseases (AD and PD)

Exclusion Criteria:

All patients for whom there are contraindications to performing MRI. Also excluded from the study will be subjects who are pregnant, or presumed to be pregnant or undergoing of lactation and subjects with claustrophobia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 patients with Alzheimer's disease (AD) and Parkinson's disease (PD)
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Development of a performant multiparametric system capable of identifying novel biomarkers of microglial polarization that can be used for diagnostic and prognostic purposes in determining the staging/progression of neurodegenerative disease | 1-36 months
  Collection and processing of multimodal imaging data and biological samples in patients with Dementia; Development of the Informatics Platform to support the interpretation of data in clinical setting

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Synlab SDN, Naples, Italy

IPD SHARING:
Plan to Share IPD: No